CLINICAL TRIAL: NCT00270374
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Hemodynamic and Clinical Effects of Natrecor (Nesiritide) Compared With Nitroglycerin Therapy for Symptomatic Decompensated CHF, The VMAC Trial: Vasodilation in the Management of Acute Congestive Heart Failure
Brief Title: A Study Comparing Blood Flow and Clinical and Safety Effects of the Addition of Natrecor (Nesiritide), Placebo or Intravenous Nitroglycerin to Standard Care for the Treatment of Worsening Congestive Heart Failure.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005206
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Symptomatic Decompensated Congestive Heart Failure; Congestive Heart Failure in Acute Coronary Syndrome
Keywords: Congestive heart failure; CHF; Left-sided heart failure; Right-sided heart failure; Systolic Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic | interventions — Natriuretic Peptide, Brain

ARMS (1):
- 001 (Experimental): nesiritide
  Interventions: Drug: nesiritide

INTERVENTIONS:
Drug: nesiritide

SUMMARY:
The purpose of this study is to compare the hemodynamic (blood flow) and clinical effects of the study drug, Natrecor (nesiritide, a recombinant form of the natural human peptide normally secreted by the heart in response to heart failure) to those of intravenous nitroglycerin or placebo, when added to the standard care therapy that is usually administered in the treatment of patients with worsening congestive heart failure.

DETAILED DESCRIPTION:
Advanced congestive heart failure (CHF) accounts for over 1 million hospital admissions yearly in the U.S. and is also associated with a high rate of readmission to the hospital within a short turn-around time period following discharge. CHF is associated with a relatively high death rate, up to 40 or 50% in 2 years. The risk of sudden cardiac death in patients with CHF is 6 to 9 times greater than that of the general population. Despite medical advances, some patients are unresponsive to the oral medications used to treat CHF and require added therapy. Such patients are typically New York Heart Association (NYHA) Class III and IV, and require intravenous (IV) therapy with inotropic agents. Inotropic agents are drugs that influence muscular contractility. IV administration with inotropic drugs requires careful patient selection and close monitoring to ensure safe and effective therapy.

There are many medical conditions that lead to worsening CHF and these underlying conditions contribute to a significant and potentially life-threatening loss of cardiac function. Some of these are conditions that lead to abnormal cardiac contraction and/or relaxation (e.g., coronary arterial disease, hypertension, diabetes, drug or alcohol toxicity); conditions that lead to volume or pressure overload (mitral or tricuspid valve regurgitation, hyperthyroidism); and conditions that limit ventricle filling (e.g., mitral or tricuspid valve stenosis). However, many patients have a condition of dilated cardiomyopathy, an abnormality of the heart muscle wall in which the walls of the heart become stretched and weakened, with no easily identifiable cause. Any risk factor may cause CHF, but combinations dramatically increase the risk of developing CHF.

Natriuretic peptides ANP and BNP are small molecules and are the group of naturally-occuring substances that act in the body to oppose the activity of the renin-angiotensin-aldosterone (RAA) system. They serve as counter-regulatory hormones and are secreted in response to the increased atrial and ventricular stretching that occurs in secondary increased blood volume. Natrecor (nesiritide) is the proprietary name for the IV formulation of human B-type natriuretic peptide (hBNP).

In-patient treatment for acutely decompensated CHF with intravenous vasodilator therapy (such as nitroglycerin or nitroprusside) is useful for a number of reasons. Vasodilators reduce ventricular filling pressure and volume, decreasing pulmonary congestion and the resulting symptoms of breathlessness. Intravenous vasodilators may also achieve afterload reduction leading to decreased mitral regurgitation and increased forward stroke volume. IV administration of externally produced hBNP leads to vasodilation, antagonism of the renin-aldosterone system and an increase in diuresis. hBNP may be a potent agent for the treatment of CHF, with a unique combination of desirable blood flow throughout the body, hormones secreted by the sympathetic nervous system, and renal effects not possessed by currently available therapies. In a 6-hour placebo-controlled comparison in patients with acutely decompensated CHF, Natrecor® was associated with significant improvements in the symptoms of CHF (including dyspnea and fatigue), a decrease in aldosterone, and an increase in urine output. (According to LeJemtel et al 1998) The VMAC trial (Vasodilation in the Management of Acute CHF) is a double-blinded, randomized, active-controlled and placebo-controlled study in which the study drug would be added to standard care therapies such as diuretics, dobutamine, or dopamine. This study compares the effects of the addition of Natrecor®, nitroglycerin, or placebo to standard care (diuretics, dobutamine, dopamine, or other long-term cardiac therapies) in patients requiring hospitalization for the treatment of dyspnea at rest due to acutely decompensated CHF. Based on the cumulative experience with Natrecor, the dose of Natrecor was modified for the VMAC trial to a 2-µg/kg bolus followed by a 0.01-µg/kg/min infusion.

The primary objective of the VMAC study is to compare the blood flow and observe treatment and safety effects of the new dose of Natrecor to placebo, when added to standard care, in the treatment of acutely worsening CHF. The primary overall outcome that the study plan is based upon are the changes from the beginning of a study to 3 hours after the start of study drug, in pulmonary capillary wedge pressure (PCWP) (in subjects who have right heart catheters only) and the subject's self-evaluation of their breathing difficulties. The secondary objective is to compare the hemodynamic, (blood flow throughout the body) and clinical effects of Natrecor® with IV nitroglycerin and placebo. Additional objectives include a comparison of the use of other IV vasoactive agents and/or IV diuretics and the effects on other hemodynamic variables. The hypothesis of this study is that using the modified dose of Natrecor, (a 2-µg/kg bolus followed by a 0.01-µg/kg/min infusion) will achieve peak effects sooner than with previously studied doses, to sustain effects for at least 48 hours, and minimize excessive effects on blood pressure. Natrecor or placebo, administered as an intravenous 2-µg/kg bolus, followed by a fixed-dose infusion of 0.01-µg/kg/min.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspnea (difficulty breathing and shortness of breath) at rest, while supine, or immediately upon minimal activity such as talking, eating, or bathing
* having evidence of heart disease, rather than pulmonary disease, as the primary cause for the dyspnea (by demonstrating at least two of the following: jugular venous distension, paroxysmal nocturnal dyspnea or 2-pillow orthopnea within 72 hours before the start of study drug, abdominal discomfort due to hepatosplanchnic congestion, chest x-ray with findings indicative of heart failure)
* having elevated cardiac filling pressures either by clinical estimate in non-catheterized patients, or a measured pulmonary capillary wedge pressure (PCWP) >= 20 mm Hg in catheterized patients
* requiring hospitalization and intravenous therapy for at least 24 hours for the treatment of acutely decompensated heart failure.

Exclusion Criteria:

* NPatients having systolic blood pressure consistently less than 90 mm Hg
* having cardiogenic shock (a sudden decrease in blood pressure that results in decreased perfusion of body tissues and organs), volume depletion, or any other clinical condition that would contraindicate the administration of an intravenous agent with potent vasodilating properties
* having their most recent pulmonary capillary wedge pressure (PCWP) < 20 mm Hg within 24 hours before randomization
* having a clinical status so acutely unstable that the potential subject could not tolerate placement of a right heart catheter or the 3-hour placebo period
* unable to have intravenous nitroglycerin withheld (e.g., intravenous nitroglycerin for management of an acute coronary syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 1999-10; Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 3 hours after the start of study drug in PCWP (pulmonary capillary wedge pressure) in subjects who have right heart catheters; Change from baseline in dyspnea (difficult breathing) 3 hours after the start study drug

SECONDARY OUTCOMES:
Effect on PCWP (pulmonary capillary wedge pressure) and dyspnea (difficult breathing) 1 hour after the start of study drug; Onset of effect on PCWP; Effect on PCWP 24 hours after the start of study drug; Overall safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Result] Publication Committee for the VMAC Investigators (Vasodilatation in the Management of Acute CHF). Intravenous nesiritide vs nitroglycerin for treatment of decompensated congestive heart failure: a randomized controlled trial. JAMA. 2002 Mar 27;287(12):1531-40. doi: 10.1001/jama.287.12.1531. PMID 11911755